CLINICAL TRIAL: NCT06750692
Title: Comparison of the Effects of Mirror Therapy,repetitive Transcranial Magnetic Stimulation and Robotic-assisted Hand Therapy Added to Neurological Rehabilitation on Upper Extremity Functions, Quality of Life and Pain in Stroke Patients
Brief Title: Comparison of the Effects of Mirror Therapy,rTMS and Robotic-assisted Hand Therapy in Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Selma Eroğlu, Associate Professor, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SBH2025
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Stroke; Upper Extremity Dysfunction; Neuropathic Pain; Quality of Life; Neurologic Disorder
Keywords: Mirror Therapy; Repetitive Transcranial Magnetic Stimulation; Hand-Finger Robot
MeSH Terms: conditions — Stroke; Neuralgia; Nervous System Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Single-Blinded Prospective Randomized Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental: Mirror therapy (Experimental): The first group of participants will receive mirror therapy for 4 weeks, 5 sessions per week for a total of 20 sessions of upper extremity mirror therapy.
  Interventions: Other: Procedure: Mirror therapy
- Experimental: Low Frequency rTMS Protocol (Experimental): The second group will receive a total of 20 sessions of Repetitive Transcranial Magnetic Stimulation (rTMS) to the contralateral M1 upper extremity motor cortex region at low frequency (1Hz) and intensity of 100%-110% of the resting motor threshold, 5 sessions per week for 4 weeks.
  Interventions: Device: Device: Low Frequency rTMS Protocol
- Experimental: Robotic-assisted hand therapy (Experimental): In the Robot Assisted Therapy group, a total of 20 sessions will be applied to the hemiplegic upper extremity with AMADEO (Tyromotion Austria) 5 days a week for 4 weeks.
  Interventions: Device: Robotic-assisted hand therapy

INTERVENTIONS:
Other: Procedure: Mirror therapy — The first group of participants will receive a total of 20 sessions of upper extremity mirror therapy program, 5 sessions per week for 4 weeks.
  Arms: Experimental: Mirror therapy
Device: Device: Low Frequency rTMS Protocol — Repetitive Transcranial Magnetic Stimulation (rTMS) will be applied at an intensity of 100-110% of the resting motor threshold and low frequency (1 Hz) to the contralateral M1 upper extremity motor cortex region for a total of 20 sessions, 5 sessions per week for 4 weeks. rTMS application is planned to provide magnetic stimulation with the stimulator of the Magventure MagPro R30 device.
  Arms: Experimental: Low Frequency rTMS Protocol
Device: Robotic-assisted hand therapy — In the Robot Assisted Therapy group, a total of 20 sessions will be applied 5 days a week for 4 weeks using continuous passive range of motion, active assistive exercise and play therapy programs for hemiplegic upper extremities with AMADEO (Tyromotion Austria).
  Arms: Experimental: Robotic-assisted hand therapy

SUMMARY:
The aim of the study is to investigate the comparison of the effects of mirror therapy, Repetitive Transcranial Magnetic Stimulation and robot-assisted hand therapy added to conventional neurological rehabilitation on upper extremity function, quality of life and pain in stroke.

DETAILED DESCRIPTION:
Stroke is the second leading cause of death in adults and an important cause of long term disability. Functional limitations that develop in the post stroke period affect participants quality of life and activities of daily living. Today, despite advances in rehabilitation and new pharmacologic strategies, stroke related upper extremity function, quality of life and pain treatment may not always achieve the desired results. There are new approaches in stroke rehabilitation such as mirror therapy, Repetitive Transcranial Magnetic Stimulation, robot-assisted hand therapy. Three groups will take part in this study. All three groups will receive a total of 20 sessions of conventional neurological rehabilitation program 5 days a week for 4 weeks. In addition to the first group, a total of 20 sessions of upper extremity mirror therapy program will be applied for 4 weeks, 5 sessions per week. The second group will receive Repetitive Transcranial Magnetic Stimulation (rTMS) to the contralateral M1 upper extremity motor cortex region at low frequency (1Hz) and at an intensity of 100%-110 of the resting motor threshold, 5 sessions per week for a total of 20 sessions for 4 weeks. The third group will receive a total of 20 sessions of robot-assisted hand therapy using AMADEO (Tyromotion Austria) 5 days a week for 4 weeks.These three groups will be compared in terms of upper extremity function, quality of life and pain.Brunstroom, Mini Mental Test, Modified Ashworth Scale, Fugl Meyer Upper Extremity Motor Assessment Scale, Box Block Test, Nine Hole Pag Test, ABILHAND Stroke Hand Function Questionnaire, Stroke Impact Questionnaire, Stroke Specific Quality of Life Scale, Visual Analog Scale , LANNS neuropathic pain assessment scale, 4 Question Neuropathic Pain Questionnaire, Beck Depression Inventory, Beck Anxiety Scale, Pittsburgh Sleep Quality Index, MEP (motor evoked potential) measurement will be done . Participants will be evaluated by a physician twice at the beginning and at the end of treatment (4th week).

ELIGIBILITY:
Inclusion Criteria:

* Patients who applied to Afyonkarahisar Health Sciences University Hospital Physical Medicine and Rehabilitation Polyclinic with the diagnosis of hemiplegia after a cerebrovascular accident in the inpatient ward or as an outpatient for neurological rehabilitation after taking the anamnesis and physical examination, who met the inclusion criteria and eliminated the exclusion criteria
* Female and male patients between the ages of 40-80
* stroke at least 3 months ago
* voluntarily agreed to participate in the study regularly, whose health status is suitable for rehabilitation and who are medically stable
* mini mental test score of 15 and above
* Neurologically stable patient

Exclusion Criteria:

* significant comorbidities such as serious heart disease (aortic stenosis, angina, hypertrophic cardiomyopathy, arrhythmia, pacemaker) and uncontrolled hypertension
* history of epilepsy, antiepileptic drug use
* intracranial metal objects
* intraauricular implants
* cognitive dysfunction
* upper extremity peripheral nerve injuries
* malignancy
* active infection
* skin infections or open wounds in the application area
* inflammatory diseases
* orthopedic injuries that may limit maximum effort capacity
* brain lesion or drug use history that may affect the seizure threshold
* increased intracranial pressure
* uncontrolled migraine
* severe spasticity in the hand (MAS≥3)
* contracture in the hand
* have had a fracture or surgery on the hemiplegic side in the last 6 months
* severe visual impairment
* severe depression

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-12-27 (Actual); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Fugl Meyer Upper Extremity Assessment Questionnaire | Baseline and Post-treatment (4th week)
  The Fugl Meyer Upper Extremity Motor Assessment Scale was developed to quantitatively assess sensorimotor recovery after stroke. It was prepared based on Brunnstrom's stages of motor recovery. The FMUE Scale consists of 33 items, each scored from 0 to 2, where 0 = cannot perform, 1 = partially performs, and 2 = fully performs. The total score is 66. A range of data is available for the minimum clinically important differences for the FMUE Scale. A change of 4 to 7 points in chronic stroke, 12 points in subacute stroke, and 9 to 10 points is considered clinically significant.Higher scores indicate better upper limb functional recovery.

SECONDARY OUTCOMES:
Brunnstrom Staging | Baseline and Post-treatment (4th week)
  It is a test that evaluates the motor development of hemiplegic participants. In this test, the neurophysiological recovery process of the hemiplegic participant is defined as 6 stages. According to this staging, the lowest stage is stage 1 (flaccid, stage without voluntary movement), and the highest stage is stage 6 (stage with isolated joint movement). In Brunnstrom staging, the hand and upper extremity are evaluated separately.
Mini Mental Test | Baseline
  It is a widely used cognitive screening test. The total score is 30 points. It has been stated that scores below 15 indicate low cognitive function, scores between 15-26 indicate medium, and scores above 26 indicate high cognitive level.
Modified Ashworth Scale | Baseline and Post-treatment (4th week)
  The modified Ashworth scale is a muscle tone assessment scale used to assess the resistance experienced during passive range of motion, which does not require any instrumentation and is quick to perform.This scale grades the muscle tone from 0 (normal) to 4 (severe spasticity). Higher scores indicating sever spasticity.
Box Block Test | Baseline and Post-treatment (4th week)
  It is used to evaluate rough manual dexterity based on performance (time). 150 small wooden cubes are filled from the box with the participant's hand to be tested into the adjacent box. The participant is asked to throw one cube at a time into the semi-empty box. How many cubes are thrown in 60 seconds is counted. The result gives the score. How many cubes are thrown in 60 seconds is counted. The result gives the score. The higher the score, the higher the success rate.
Nine Hole Peg Test | Baseline and Post-treatment (4th week)
  This test measures dexterity based on performance (in seconds). A wooden board with nine holes on it, 9 short wooden sticks and a box in which the wooden sticks can be placed are placed in front of the participant. Using the hand to be evaluated, the participant is asked to place the wooden sticks in the box into the holes on the panel as quickly as possible. Then, he is asked to put the sticks back into the box one by one. The completion time of the test is determined by a stopwatch. In this test, which evaluates manual dexterity based on performance, the success rate increases as the time gets short
Pittsburgh Sleep Quality Index (PSQI) | Baseline and Post-treatment (4th week)
  The Pittsburgh Sleep Quality Index (PSQI) is an 18 item questionnaire that assesses sleep quality and disturbances over the past month. The investigators will use the 3-factor scoring, which has been shown to have superior psychometric properties. The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality
ABILHAND Stroke Hand Function Questionnaire | Baseline and Post-treatment (4th week)
  The ABILHAND Hand Questionnaire was developed in 1998 to measure participant perceived dexterity. It contains 23 questions about how difficult the participant has to do the activities. impossible (0 points), difficult (1 point), easily (2 points) options is marked. The total score is 46.Higher scores indicate better hand functional recovery.
Stroke Impact Scale | Baseline and Post-treatment (4th week)
  The Stroke Impact Scale (SIS) is a stroke specific health status measure. It consists of a total of 59 items and 8 sections. The participant is asked to evaluate the difficulty experienced in completing each item in the last week on a five point Likert scale. A score of one indicates that the participant could not complete the item, and a score of five indicates that the participant had no difficulty in completing it. It also includes a visual analog scale (0: No improvement, 100: Complete recovery) regarding the general perception of recovery after stroke.
Stroke Specific Quality of Life Scale | Baseline and Post-treatment (4th week)
  Specific Quality Of Life scale (SSQOL) is a participant centered outcome measure intended to provide an assessment of health related quality of life specific to participants with stroke. The original test consists of 49 items encompassing 12 domains. Each item is ranked on a 5 point scale, with higher scores indicating better function.
The Self Assessment of Neuropathic Symptoms and Signs (S-LANSS) | Baseline and Post-treatment (4th week)
  The SLANSS scale is a scale that helps to distinguish neuropathic pain from nociceptive pain. Unlike the LANSS scale, the physician does not examine the participant in this scale, so it is easier to administer. The S-LANSS scale consists of a total of 7 questions. The participant fills in this scale on his/her own. The first 5 questions ask about pain symptoms, while the last 2 questions include the participant's self administered clinical examination. The answers to the questions are yes/no. Each question has a different score. The total score on the scale is 24. A total score of 12 or more indicates neuropathic pain.
Beck Depression Scale | Baseline and Post-treatment (4th week)
  The Beck Depression Scale is a 21 item self report inventory designed to assess the presence and severity in depressive symptoms. Each item is rated on a 4-point Likert type scale ranging from 0 to 3, based on the severity in the last two weeks. Higher scores indicating worse level of depression.
Beck Anxiety Inventory | Baseline and Post-treatment (4th week)
  The anxiety level of the participants was assessed using the Beck Anxiety Inventory (BAI). BAI is used to determine the severity of anxiety symptoms experienced by individuals. It is a Likert type scale with 21 headings that participants themselves score between 0-3, the score that can be obtained varies between 0-63, and the higher the score, the greater the anxiety experienced by the individual.
Neuropathic Pain Questionnaire in 4 Questions | Baseline and Post-treatment (4th week)
  ''Neuropathic Pain Questionnaire in 4 Questions'' is a short form designed to detect and diagnose neuropathic pain symptoms. The questionnaire consists of 10 questions to assess the symptoms experienced by the participant. These questions question signs and symptoms specific to neuropathic pain. A score between 0 and 10 is determined.
Visual Analog Scale (VAS) | Baseline and Post-treatment (4th week)
  The participant' musculoskeletal pain severity was assessed with the visual analog scale (VAS). The meanings of the numbers placed from 0 to 10 on a 10 cm line were explained to the participants. It was explained that no pain was 0, the most severe pain felt in life was 10, and moderate pain was 5 points. According to these explanations, the participants were asked to score their pain levels considering the last week.
Neurophysiological Measurements | Baseline and Post-treatment (4th week)
  Neurophysiologic evaluations of all participants will be performed twice before and 4 weeks after treatment. Participants will undergo MEP (motor evoked potential) measurement with TMS stimulation. The MagVenture MagPro R30 (Denmark) transcranial magnetic stimulation device in the Neuromodulation Unit will be used with Figure Eight Coil.

CONTACTS AND LOCATIONS:
Overall Officials: Selma Eroglu, MD, Principal Investigator — Afyonkarahisar Health Sciences University
Locations (1):
- Afyonkarahisar Health Sciences University, Afyonkarahisar, Turkey (Türkiye)

REFERENCES:
- [Background] Suganuma Y, Shimode C, Yamamoto H. Conjugation in Tetrahymena: formation of a special junction area for conjugation during the co-stimulation period. J Electron Microsc (Tokyo). 1984;33(1):10-8. No abstract available. PMID 6491567
- [Background] Jia F, Zhao Y, Wang Z, Chen J, Lu S, Zhang M. Effect of Graded Motor Imagery Combined With Repetitive Transcranial Magnetic Stimulation on Upper Extremity Motor Function in Stroke Patients: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2024 May;105(5):819-825. doi: 10.1016/j.apmr.2023.12.002. Epub 2023 Dec 17. PMID 38110138
- [Background] The presidents. Frank Abbott, 1887-1888. J Am Dent Assoc. 1981 Apr;102(4):471. No abstract available. PMID 7012218